CLINICAL TRIAL: NCT04053062
Title: A Phase I Study to Evaluate the Safety and Efficacy of PSMA-CART Co-expressing LIGHT in Treating Patients With Castrate-Resistant Prostate Cancer (CRPC)
Brief Title: LIGHT-PSMA-CART in Treating Patients With Castrate-Resistant Prostate Cancer
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to efficacy evaluation
Sponsor: Bioray Laboratories (Industry)
Collaborators: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-CAR-00CH1
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Castrate-Resistant Prostate Cancer
Keywords: Castrate-Resistant

STUDY DESIGN:
Intervention Model Description: 3 x 10^6/ KgBW; 6 x 10^6/ KgBW
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LIGHT-PSMA-CART (Experimental): Patients undergo leukapheresis. Patients then receive cyclophosphamide and fludarabine on days -6 to -4. Patients receive LIGH-PSMA-CART IV at split doses from day 0 on.
  Interventions: Biological: LIGHT-PSMA-CART cells

INTERVENTIONS:
Biological: LIGHT-PSMA-CART cells — LIGHT-PSMA-CART cells will be given IV at split doses
  Other Names: Autologous PSMA-specific chimeric antigen cells co-expressing LIGHT

SUMMARY:
This is a single center, single arm Phase I study to establish the safety and efficacy of intravenously administered lentivirally transduced LIGHT-PSMA-specific CAR modified autologous T cells (PSMA-CART cells) in patients with CRPC.

DETAILED DESCRIPTION:
This is a Phase I study evaluating the safety and efficacy of PSMA targeting autologous CAR T cells co-expressing LIGHT in a 3+3 dose escalation design. Cohort 1 subjects (N=3 or 6) will receive a tolal dose of 3x 10^6/kg body weight (KgBW) LIGHT-PSMA-CART cells at split doses after a conditioning chemotherapeutic regimen(Cy+Flu). If 1 DLT/3 subjects occurs, the study will enroll an additional 3 subjects at this dose level. If 0 DLT/3 subjects or 1 DLT/6 subjects occurs, the study will advance to Cohort 2, with a total dose of 6 x 10^6/ KgBW.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand and voluntarily sign informed consent.
* Male, aged 18 to 75 years old.
* Expected survival > 6 months.
* CRPC patients: Prostate cancer is still progressing after continuous androgen deprivation therapy. Including, castrate levels of serum testosterone (<50ng/dl or <1.7nmol/L); or prostate specific antigen (PSA) increased more than 50% at intervals of one week or three consecutive times, and PSA>1 ug/L; or imaging scans revealed two or more new lesions or enlargement of soft tissue lesions that met the criteria for evaluating solid tumor response.
* CRPC patients received abiraterone or chemotherapy for 3 months or more, and were ineffective or progressive (PSA continued to rise for 3 months, or bone scan/whole-body MRI/PET-CT showed local recurrence or new metastasis).
* Immunohistochemical staining of repetitive biopsy tissues showed the expression of PSMA in tumor cells was more than 50%.
* ECOG score <2.
* Hgb > 10 g/dl.
* PLT > 100×109/L.
* ANC > 1.5×109/L.

Exclusion Criteria: Subjects who meet any of the following exclusion criteria will be excluded

* Prior treatment with any immunotherapy, including CART therapy, tumor vaccine therapy, radium-223, checkpoint inhibitors.
* Prior treatment with any PSMA targeting therapy.
* Subjects with severe mental disorders.
* Subjects with severe cardiovascular diseases: a, New York Heart Association (NYHA) stage III or IV congestive heart failure; b, history of myocardial infarction or coronary artery bypass grafting (CABG) within 6 months; c, clinical significance of ventricular arrhythmia, or history of unexplained syncope, non-vasovagal or dehydration; d, history of severe non-ischemic cardiomyopathy; e, the left ventricular ejection fraction (LVEF < 55%) was decreased by echocardiography or MUGA scan (within 8 weeks before PBMC collection), and abnormal interventricular septal thickness and atrioventricular size associated with myocardial amyloidosis.
* Patients with ongoing or active infection.
* Aspartate aminotransferase or Alanine aminotransferase >2.5*ULN; CK>1.5*ULN; CK-MB>1.5*ULN; TnT>1.5*ULN.
* Total bilirubin >1.5*ULN.
* Partial prothrombin time or activated partial thromboplastin time or international standardized ratio > 1.5*ULN without anticoagulant treatment.
* History of participation in other clinical studies within 3 months or treatment with any gene therapy product.
* Intolerant or allergic to cyclophosphamide or fludarabine.
* Subjects not appropriate to participate in this clinical study judged by investigators.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | 28 days
  All adverse events (AEs) will be listed and summarized. Summaries of laboratory data will include, at a minimum, treatment-emergent laboratory abnormalities. Summaries of AEs and laboratory abnormalities will be based on the All Treated analysis set.

SECONDARY OUTCOMES:
PSA response rate | 24 weeks
  proportion of patients with ≥50% PSA decline from baseline at any time point after therapy and maintained for ≥4 weeks
Radiographic response rate by RECIST 1.1 & PCWG3. | 24 weeks
  Proportion of patients with a best response of either complete response or partial response, assessed using Prostate Cancer Working group3(PCWG3) response criteria &RECIST 1.1.
Duration time of CART cells in vivo | 24 weeks
  Number of persistent PSMA-CART cells detected by Q-PCR or flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Shancheng Ren, Professor, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China